CLINICAL TRIAL: NCT06973356
Title: An Exploratory Clinical Study of Anti-CD19/BCMA CAR Gene Vector Injection (LCAR1901) for the Treatment of Relapsed and Refractory Immune Thrombocytopenia
Brief Title: Anti CD19/BCMA CAR Gene Therapy for Relapsed/Refractory Immune Thrombocytopenia
Acronym: LCAR1901
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SWKCART25032401
Record Dates: First submitted 2025-05-06; First posted 2025-05-15 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: immune thrombocytopenia; Autoimmune diseases
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Anti-CD19/BCMA CAR gene vector injection (Experimental): Arm Description: Intravenous infusion of Anti-CD19/BCMA CAR gene vector injection
  Interventions: Drug: Anti-CD19/BCMA CAR gene vector injection will be injected intravenously on a one-time basis.

INTERVENTIONS:
Drug: Anti-CD19/BCMA CAR gene vector injection will be injected intravenously on a one-time basis. — Description: A single intravenous infusion of anti-CD19/BCMA CAR gene vector injection(dose-escalating infusion of 1.0-4.0 x10^6 TU/kg）.

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 18 participants with treatment of relapsed and refractory immune thrombocytopenia. This study aims to evaluate the safety and efficacy of the treatment with an Anti- CD19/BCMA CAR gene vector injection

ELIGIBILITY:
Inclusion Criteria:

* 1. Age≥ 18 years old, regardless of gender. 2. Clinical diagnosis of primary immune thrombocytopenia for at least 6 months, platelet count < 30×10^9/L within 48 hours before participating in the study.

  3. Positive anti-platelet glycoprotein autoantibodies (such as GPIIb/IIIa). 4. Prior second-line ITP therapy (first-line treatment includes: corticosteroids or immunoglobulins; Second-line therapies include thrombopoietin receptor agonists (eg, eltrombopag, romiplostim) and/or rituximab, but are ineffective (platelet count < 30×10^9/L after treatment, or platelet count does not increase twice as much as baseline, or there is bleeding), or relapse after effective treatment (platelet count falls below 30×109/L after effective treatment, or falls below baseline, or bleeding symptoms) or is difficult to maintain after discontinuation of TPO agonists.

  5. Bone marrow examination shows megakaryocytosis or normal. 6. Basic normal functions of important organs:Echocardiography shows an ejection fraction of ≥50% and no significant abnormalities on ECG.Creatinine clearance (CrCl) (Cockcroft-Gault formula) ≥ 30 mL/min.Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × upper limit of normal (ULN).Total bilirubin (TBIL) and alkaline phosphatase (AKP or ALP) ≤ 2.0× ULN (Gilbert's syndrome ≤3.0×ULN).Absolute lymphocyte count (ALC) ≥ 0.5×10^9/L; Absolute neutrophil count (ANC) ≥1×10^9/L; Hemoglobin (Hb) ≥ 60 g/L; Platelet count ≥ 10×10^9/L.Oxygen saturation > 92%.ECOG performance status ≤2 7. Males and women of childbearing potential must agree to use effective contraception from the time of signing the informed consent form until 1 year after the use of the study drug. Women of childbearing potential must have a negative blood pregnancy test at screening and prior to drug infusion and must not be breastfeeding.

Exclusion Criteria:

* 1. Thrombocytopenia caused by myelodysplastic syndrome, early aplastic anemia, atypical aplastic anemia, thrombotic thrombocytopenic purpura, etc.

  2. During the screening period, bone marrow examination showed myelofibrosis MF≥2 (European consensus scoring standard Thieleja 2005) or bone marrow examination showed the presence of a primary disease other than ITP that can lead to thrombocytopenia.

  3. History of hypersensitivity to any component of the therapeutic medication. 4. Major organs: NYHA class III to IV congestive heart failure. Myocardial infarction or coronary artery bypass grafting (CABG) or coronary artery stent implantation within 6 months. Ventricular arrhythmias, or history of unexplained syncope (excluding vasovagal syncope or dehydration). History of severe non-ischemic cardiomyopathy.

  5. Malignant disease within 3 years prior to screening, except for the following: malignant disease that has been curatively treated before enrollment and has no known active disease for 3 years ≥; or well-treated non-melanoma skin cancer with no evidence of disease.

  6. Symptomatic deep vein thrombosis or pulmonary embolism within the past 6 months or currently requiring anticoagulation.

  7. Participated in other interventional clinical studies within 1 month prior to screening.

  8. Vaccination of live attenuated vaccine within 4 weeks prior to screening. 9. Stroke or seizure within 6 months prior to signing the ICF (excluding old lacunar cerebral infarction).

  10. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titer test exceeds the normal range; Hepatitis C virus (HCV) antibody is positive and the hepatitis C virus (HCV) RNA titer in peripheral blood exceeds the normal range; positive for human immunodeficiency virus (HIV) antibodies; Positive syphilis test.

  11. Known history of bone marrow stem cell disease 12. Other conditions that the investigators consider unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-16 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
1. Adverse events | up to 1 years
  Total number, incidence and severity of adverse events (AEs) in patients of LCAR1901 infusion. The AEs will be assessed according to the 2019 Consensus on Cytokine Release Syndrome and Immune-cell-associated Neurotoxicity published by the American Society of Transplantation and Cell Therapy (ASTCT), the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 and EBMT 2019 consensus

SECONDARY OUTCOMES:
2. The persistence of CAR gene vector injection | up to 1 years
  Assessing the trafficking of CAR gene vector injection in the peripheral blood at the time of each infusion as well as at each time of follow-up by flow cytometry. Peripheral blood will be collected prior to the initial infusion and will be set as baseline
Overall remission rate | up to 1 years
  Complete response (CR): Platelet count ≥ 100 × 10^9/L and no bleeding; Partial response (PR): platelet count<100 × 10^9/L, but increased by at least 2 times compared to baseline platelet count, with no bleeding symptoms

CONTACTS AND LOCATIONS:
Overall Officials: bing xing wang, M.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China; cheng chang zheng, M.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- Hunan Siweikang Therapeutic Co.Ltd, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes